CLINICAL TRIAL: NCT03739879
Title: Effectivity of Inspiratory Muscle Trainer in the Chronic Obstructive Pulmonary Disease Rehabilitation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Fariz Nurwidya, Lecturer, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: COPD Muscle Trainer
Record Dates: First submitted 2018-11-06; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Inspiratory muscle trainer; Pulmonary rehabilitation; COPD; St George Respiratory Questionnaire; 6-minute Walking Test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Patients underwent an interview about their medical history, tested spirometry using Carefusion®, and the inspiratory muscle strength was assessed using Micro RPM Carefusion®. The St George Respiratory Questionnaire (SGRQ) was used to assess the health status and the 6-minute Walking Test (6MWT) was conducted to assess functional capacity. Subject exercised using inspiratory muscle trainer (Philips Respironic®) for eight weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Inspiratory muscle training (IMT) (Experimental): Subjects exercised using inspiratory muscle trainer (Philips Respironic®) for 8 weeks. Training dose with IMT was determined by inspiratory muscle strength result and adjusted in every evaluation visit. The subject was expected to do exercise twice daily for 15 minutes each session with 30-70% intensity from determined MIP score. Exercise is monitored and noted in a logbook.
  Interventions: Device: Inspiratory Muscle Trainer Philips Respironics

INTERVENTIONS:
Device: Inspiratory Muscle Trainer Philips Respironics — Subjects exercised using inspiratory muscle trainer (Philips Respironic®) for 8 weeks. Training dose with IMT was determined by inspiratory muscle strength result and adjusted in every evaluation visit. The subject was expected to do exercise twice daily for 15 minutes each session with 30-70% intensity from determined MIP score. Exercise is monitored and noted in a logbook.

SUMMARY:
This study aimed to reveal the role of inspiratory muscles exercise using Inspiratory Muscle Trainer (IMT), which is a form of weight training. The pre- and post study of this experiment were conducted in chronic obstructive pulmonary disease (COPD) outpatient clinic during the period of September 2017 until April 2018. Patients were recruited by consecutive sampling. Inclusion criteria were stable COPD patient with The Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria A-D, who has never received prior exercise for pulmonary rehabilitation, and willing to participate in the study. The exclusion criteria included any problem with extremities and cardiovascular disease. Patients underwent an interview about their medical history, tested spirometry using CareFusion®, and the inspiratory muscle strength was assessed using Micro RPM CareFusion®. The St George Respiratory Questionnaire (SGRQ) was used to assess the health status and the 6-Minute Walking Test (6MWT) was conducted to assess functional capacity. Subject exercised using inspiratory muscle trainer (Philips Respironic®) for eight weeks.

DETAILED DESCRIPTION:
Intervention is given using Inspiratory Muscle Trainer Philips Respironic®. Impact on inspiratory muscles strength, health status, and functional capacity are observed. Muscle strength is evaluated using Micro RPM (Respiratory Pressure Meter) Carefusion®. Health status is evaluated using St. George's Respiratory Questionnaire (SGRQ), while functional capacity is evaluated by the 6-Minute Walk Test (6MWT).

Patients were recruited by consecutive sampling. This study was granted ethical approval from the Institutional Review Board (IRB) of the Faculty of Medicine Universitas Indonesia Subjects exercised using inspiratory muscle trainer (Philips Respironic®) for 8 weeks. Inspiratory muscles strength (Maximal Inspiratory Pressure, MIP) and 6MWT were done at the beginning for basic data and were re-evaluated during the second, fourth, sixth and eighth week (last week). Questionnaire (SGRQ) was done at the initial and end of research.

Training dose with IMT was determined by inspiratory muscle strength result and adjusted in every evaluation visit. The subject was expected to do exercise twice daily for 15 minutes each session with 30-70% intensity from determined MIP score. Exercise is monitored and noted in a logbook.

ELIGIBILITY:
Inclusion Criteria:

* stable COPD patient with GOLD criteria A-D,
* never got exercise for pulmonary rehabilitation before,
* willing to participate in the study by signing the written informed consent.

Exclusion Criteria:

* any problem with extremities,
* cardiovascular disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscles strength | Eighth week
  This outcome was determined by maximal inspiratory pressure (MIP)
Functional capacity | Eighth week
  This outcome was determined by 6-minutes walking test
Health status | Eighth week
  Health status was evaluated using St George Respiratory Questionnaire (SGRQ) SGRQ was a questionnaire designed to measure health impairment in asthmatic and COPD patients. It consists of three parts. First part is symptom, followed by activity and impact. Every question has its own score. The least is zero and the highest is 100. Score is calculated by dividing total score with maximum score for that component and translated into percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient COPD Clinic of Dr. Cipto Mangunkusumo Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No